CLINICAL TRIAL: NCT03109392
Title: A Randomized-controlled Trial to Compare the Effectiveness of 4% Nebulized Lignocaine Versus 10% Lignocaine Spray in Patients Undergoing Flexible Bronchoscopy
Brief Title: A Randomized Trial of 4% Nebulized Lignocaine vs. 10% Lignocaine Spray in Patients Undergoing Flexible Bronchoscopy
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Responsible Party: Principal Investigator, Ritesh Agarwal, Consultant, Department of Pulmonary Medicine, Principal Investigator, Clinical Professor, Post Graduate Institute of Medical Education and Research, Chandigarh
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: Pulm.Med/2017/001
Record Dates: First submitted 2017-03-29; First posted 2017-04-12 (Actual); Last update posted 2021-02-23 (Actual); Status verified 2021-02

CONDITIONS: Patients With Indication for Flexible Bronchoscopy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Nebulized lignocaine (Experimental): 2.5 ml of 4% lignocaine will be administered via nebulization prior to bronchoscopy
  Interventions: Drug: Nebulized Lignocaine
- Lignocaine spray (Experimental): 10 puffs of 10% (10mg/puff) lignocaine spray will be sprayed at 10 seconds intervals into the pharynx immediately prior to bronchoscopy
  Interventions: Drug: Lignocaine spray
- Combined spray and nebulization (Active Comparator): Combination of 2.5 ml of 4% lignocaine via nebulization prior to bronchoscopy and 2 puffs of 10% (10mg/puff) lignocaine spray sprayed at 10 seconds intervals into the pharynx immediately prior to bronchoscopy
  Interventions: Drug: Combined spray and nebulization

INTERVENTIONS:
Drug: Nebulized Lignocaine — 2.5 ml of 4% lignocaine will be administered via nebulization prior to bronchoscopy
  Arms: Nebulized lignocaine
Drug: Lignocaine spray — 10 puffs of 10% (10mg/puff) lignocaine spray will be sprayed at 10 seconds intervals into the pharynx immediately prior to bronchoscopy
  Arms: Lignocaine spray
Drug: Combined spray and nebulization — Combination of 2.5 ml of 4% lignocaine via nebulization prior to bronchoscopy and 2 puffs of 10% (10mg/puff) lignocaine spray sprayed at 10 seconds intervals into the pharynx immediately prior to bronchoscopy
  Arms: Combined spray and nebulization

SUMMARY:
Flexible bronchoscopy is common procedure used in the diagnosis and treatment of a variety of tracheobronchial diseases. During routine diagnostic flexible bronchoscopy, the most distressing symptom experienced by the patients is a cough, and control of a cough is vital for a successful procedure. The investigators hypothesized that either nebulized lignocaine or lignocaine spray given alone prior to flexible bronchoscopy for inducing topical anesthesia will have similar efficacy compared to the combination of the two agents.

DETAILED DESCRIPTION:
Flexible bronchoscopy is common procedure used in the diagnosis and treatment of a variety of tracheobronchial diseases. The bronchoscope can be used to sample material not only from the visualized regions but also from the more distal pulmonary parenchyma. It is a safe outpatient exam that carries little risk. While performing the procedure most of the patients express some fear of pain, difficulty in breathing, nasopharyngeal irritation, and cough. During routine diagnostic flexible bronchoscopy, the most distressing symptom experienced by the patients is a cough, and control of a cough is vital for a successful procedure. Administration of a topical anaesthetic drug to the upper airway, larynx, and tracheobronchial tree can reduce a cough and patient's discomfort. The most commonly used topical anaesthetic agent in bronchoscopy is lignocaine because of its quick onset and short duration of action with decreased toxicity as compared to other agents. There are several ways to achieve topical anaesthesia in flexible bronchoscopy including nebulization, direct spray, by tracheal injection, or via nasal, or "spray as you go" technique through the working channel of the bronchoscope. The use of topical anaesthesia, sedation, and analgesia during flexible bronchoscopy varies according to physicians, institutions and geographic locations in the world. Generally, moderate sedation is used in bronchoscopy in which patients can respond to verbal commands. Deep sedation is less commonly used in which patients cannot be easily aroused but respond to repeated or painful stimulation.

Antoniades et al. demonstrated that topical lidocaine through the bronchoscope significantly decreased cough frequency and the total dose of sedation required during flexible bronchoscopy. In a randomized controlled trial of 54 patients, Keane et al. concluded that nebulized and sprayed lignocaine have similar efficacy as topical anaesthetics in fiberoptic bronchoscopy but patients preferred the nebulized route. Noitasaeng et.al. concluded in their study that spraying lidocaine took less time to start the procedure, with greater ease of instrumentation, less incidence of hypersecretion, less gag reflex, and smooth operation during the procedure but patients preferred nebulized lidocaine administration.

At the investigators' center, it has been a routine practice to perform flexible bronchoscopy without sedation in patients who require only diagnostic flexible bronchoscopy and assessment of airway anatomy and other routine procedures such as endobronchial biopsy or transbronchial biopsy. Previously, the investigators had shown that 1% lignocaine given by spray-as-you-go method was similar in efficacy to 2% lignocaine for topical anesthesia during routine flexible bronchoscopy. However, in this study both the groups received nebulized lignocaine and lignocaine spray prior to flexible bronchoscopy in addition to lignocaine solution ad lib.

The investigators hypothesized that either nebulized lignocaine or lignocaine spray given alone prior to flexible bronchoscopy for inducing topical anesthesia will have similar efficacy compared to the combination of the two agents.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Willing for flexible bronchoscopy procedure a

Exclusion Criteria:

* Requirement of intravenous sedation to undergo any procedure including EBUS-TBNA, conventional TBNA, radial EBUS procedure and interventional pulmonary procedures
* Sensitivity to lignocaine
* Hemodynamically unstable patients (SBP < 90 mm Hg)
* Baseline hypoxemia (SpO2 <92% on room air)
* Pregnancy
* Comorbid illness such as heart failure, CKD, chronic liver disease and others
* Failure to provide informed consent

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1050 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
Patient-rated intensity of cough on a visual analog scale (VAS) | One hour
  The cough VAS is a 100-mm scale anchored by no cough on one end and worst cough on the other; the patient will indicate the severity of a cough by marking a line.

SECONDARY OUTCOMES:
Pain assessment by the patient using the faces pain rating scale | One hour
  The Wong-Baker Faces Pain Scale combines the pictures and numbers to allow pain to be rated by the user. The faces range from smiling face to a sad, crying face. A numerical rating is assigned to each face, of which there is 6 total, where zero rating means no pain with smiling face and 10 mean worst pain with crying face
Patient-rated VAS of overall satisfaction of the procedure | One hour
  VAS on a 100-mm scale
Operator-rated intensity of cough on a VAS | Immediately following the procedure
  VAS on a 100-mm scale
Total lignocaine dose | Immediately following the procedure
  Total dose of lignocaine in milligrams
Changes in respiratory rate following the procedure | Baseline and 5 minutes after the procedure
  Respiratory rate at baseline and 5 minutes after the procedure
Changes in heart rate following the procedure | Baseline, during and 5 minutes after the procedure
  Heart rate at baseline, during and 5 minutes after the procedure
Changes in blood pressure following the procedure | Baseline and 5 minutes after the procedure
  Blood pressure at baseline and 5 minutes after the procedure
Changes in oxygenation status following the procedure | Baseline, during and 5 minutes after the procedure
  Pulse oximetric saturation at baseline, during and 5 minutes after the procedure
Duration of procedure (in minutes) | Immediately following the completion of flexible bronchoscopy
  The total duration of bronchoscopy procedure in minutes
Willingness of the patient to undergo the procedure yet again, if required | One hour
  Patient will indicate the willingness to undergo the procedure again, if required by a simple yes or no
Adverse reactions related to lignocaine | One hour
  Arrhythmia, involuntary movements, convulsions, anaphylaxis and bronchospasm

CONTACTS AND LOCATIONS:
Locations (1):
- Bronchoscopy suite, PGIMER, Chandigarh, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dhooria S, Chaudhary S, Ram B, Sehgal IS, Muthu V, Prasad KT, Aggarwal AN, Agarwal R. A Randomized Trial of Nebulized Lignocaine, Lignocaine Spray, or Their Combination for Topical Anesthesia During Diagnostic Flexible Bronchoscopy. Chest. 2020 Jan;157(1):198-204. doi: 10.1016/j.chest.2019.06.018. Epub 2019 Jul 9. PMID 31299247